CLINICAL TRIAL: NCT05434013
Title: The Impact of Cigarillo Warnings on Purchasing Behaviors Among Young Adult Cigarillo Users
Brief Title: The Impact of Cigarillo Warnings on Purchasing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Brown University (Other); National Institutes of Health (NIH) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); National Cancer Institute (NCI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NE-1; R01CA260460 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Cigar Smoking
Keywords: Cigarillo smoking; Cigarillo packaging warnings
MeSH Terms: conditions — Cigar Smoking

STUDY DESIGN:
Intervention Model Description: The study will conduct a three-group, between-subjects experiment to compare varying cigarillo warning formats: Surgeon General text-only, FDA-proposed text-only, and study developed pictorial cigarillo warning labels.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of 3 conditions. In each of these conditions participants will see one of the following warning label formats on the cigarillos when they are shopping for tobacco products: a pictorial warning, a text-based warning, or a surgeon general warning. Participants don't know which condition they're assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cigarillo warnings-Surgeon General Text-Only (Experimental): Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the Surgeon General Text-Only format.
  Interventions: Behavioral: Cigarillo warnings-Surgeon General Text-Only
- Cigarillo warnings-FDA proposed text-only (Experimental): Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the FDA Proposed Text-Only format.
  Interventions: Behavioral: Cigarillo warnings-FDA proposed text-only
- Cigarillo warnings-Pictorial (Experimental): Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the Pictorial format.
  Interventions: Behavioral: Cigarillo warnings-Pictorial

INTERVENTIONS:
Behavioral: Cigarillo warnings-Surgeon General Text-Only — Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the Surgeon General Text-Only format.
  Arms: Cigarillo warnings-Surgeon General Text-Only
Behavioral: Cigarillo warnings-FDA proposed text-only — Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the FDA Proposed Text-Only format.
  Arms: Cigarillo warnings-FDA proposed text-only
Behavioral: Cigarillo warnings-Pictorial — Participants will complete 6 mock shopping trips in the Experimental Tobacco Marketplace, and be asked to spend their weekly tobacco budget. Cigarillos in the Marketplace will have one of three cigarillo warnings in the Pictorial format.
  Arms: Cigarillo warnings-Pictorial

SUMMARY:
The purpose of this study is to determine whether different cigarillo warning formats (pictorial, FDA-proposed text-only, current Surgeon General text-only) reduces demand for cigarillos. A previous study has identified that pictorial cigarillo warnings are perceived as more effective, but more information is needed on their impact. This study will address this issue by randomizing participants to see different cigarillo warning formats on cigarillo products within an online experimental tobacco marketplace. Participants will be cigarillo users who are ages 21-35.

DETAILED DESCRIPTION:
Warning labels on tobacco products convey the health risks and discourage use. Warnings are even more effective when they contain images that depict the health consequences. However, little is known about the impact of cigarillo warnings, including pictorial warnings, on consumer behavior. The Experimental Tobacco Marketplace (ETM) task examines the effects of regulations on tobacco purchasing in the context of a complex tobacco marketplace. This project aims to address the gap in the knowledge about cigarillo risk communication by providing information on best practices for cigarillo warnings. Identifying effective cigarillo warnings is important to inform policy and guide research on effectively communicating risk to ultimately decrease use and tobacco-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarillo users: used cigarillos at least one time per week in the past month
* Members of the Kantar Media panel

Exclusion Criteria:

* Non-English speakers
* Non-current cigarillo users
* Not members of Kantar Media

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1578 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Ross, PhD, Principal Investigator — BU School of Public Health
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data may be provided to qualified investigators starting 9 months and ending 36 months after publication. Investigators proposing to use the data must receive a data use agree with Wake Forest University Health Sciences and seek approval from an Institutional Review Board (IRB), or similar body identified for this purpose.
Supporting Information: SAP, ICF
Time Frame: 9-36 months following publication
Access Criteria: Qualified researchers engaged in independent scientific research with IRB approval and a data use agreement with Wake Forest University Health Sciences.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Started | 526 | 526 | 526
Completed | 526 | 526 | 526
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial | Total
Number analyzed (Participants) | 526 | 526 | 526 | 1578
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (4.1) | 28.8 (4.3) | 28.9 (4.3) | 28.9 (4.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity
  Participants
    Female | 283 | 294 | 301 | 878
    Male | 235 | 226 | 219 | 680
    Unknown/Not Reported | 8 | 6 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 49 | 52 | 155
  Not Hispanic or Latino | 469 | 475 | 471 | 1415
  Unknown or Not Reported | 3 | 2 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 2 | 9
  Asian | 4 | 8 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 262 | 266 | 259 | 787
  White | 202 | 196 | 201 | 599
  More than one race | 24 | 28 | 24 | 76
  Unknown or Not Reported | 29 | 24 | 32 | 85
Region of Enrollment [Number; unit: participants]
  United States | 526 | 526 | 526 | 1578

OUTCOME MEASURES:

1. Primary Outcome: Average Total Number of Cigarillos Purchased
Description: Participants in each arm will participate in six mock shopping trips with a specified budget. They will purchase (mock) single cigarillos. The primary outcome is the average number of cigarillos purchased during each of the six mock shopping trips.
Time Frame: Within the 20-minute survey
Measure: Mean (Standard Deviation); unit: cigarillos
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 446 | 428 | 428
cigarillos
  Cigarillo price $0.25 | 6.33 (11.20) | 6.28 (9.75) | 6.64 (10.01)
  Cigarillo price $0.50 | 4.98 (7.91) | 6.45 (12.44) | 6.14 (10.09)
  Cigarillo price $0.75 | 4.36 (7.08) | 5.29 (10.83) | 4.66 (7.40)
  Cigarillo price $1.50 | 2.81 (4.28) | 3.66 (6.96) | 3.09 (4.38)
  Cigarillo price $3 | 1.82 (3.01) | 2.19 (3.83) | 1.96 (2.81)
  Cigarillo price $6 | 1.00 (1.62) | 1.14 (1.95) | 1.04 (1.77)

2. Secondary Outcome: Average Total Amount of mg Combusted Tobacco Purchased
Description: Participants will participate in six mock shopping trips with a specified budget. They will have the option to purchase (mock) tobacco products in addition to cigarillos: cigarettes, menthol cigarettes, e-cigarettes/vaping devices, oral nicotine. This outcome will be the sum mg of the number of combusted non-cigarillo tobacco products purchased during each of the six mock shopping trips
Time Frame: Within the 20-minute survey
Measure: Mean (Standard Error); unit: mg of combusted tobacco purchased
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 446 | 428 | 428
mg of combusted tobacco purchased
  Shopping Trip 1 | 445.06 (46.29) | 404.52 (30.56) | 395.66 (27.59)
  Shopping Trip 2 | 339.39 (27.34) | 416.61 (34.95) | 401.25 (38.88)
  Shopping Trip 3 | 296.12 (24.37) | 363.16 (33.61) | 360.90 (33.81)
  Shopping Trip 4 | 230.15 (20.73) | 274.97 (23.35) | 277.28 (29.80)
  Shopping Trip 5 | 181.61 (18.50) | 213.83 (20.12) | 219.56 (28.03)
  Shopping Trip 6 | 160.71 (18.30) | 171.90 (18.60) | 168.82 (19.88)

3. Secondary Outcome: Average Total Amount of mg Non-combusted Tobacco Purchased
Description: Participants will participate in six mock shopping trips with a specified budget. They will have the option to purchase (mock) tobacco products in addition to cigarillos: cigarettes, menthol cigarettes, e-cigarettes/vaping devices, oral nicotine. This outcome will be the sum mg of the number of non-combusted tobacco products purchased during each of the six mock shopping trips.
Time Frame: Within the 20-minute survey
Measure: Mean (Standard Error); unit: mg of non-combusted tobacco purchased
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 446 | 428 | 428
mg of non-combusted tobacco purchased
  Shopping Trip 1 | 134.81 (17.75) | 133.72 (18.23) | 148.93 (20.12)
  Shopping Trip 2 | 106.68 (11.19) | 122.98 (22.81) | 126.93 (17.02)
  Shopping Trip 3 | 120.26 (18.11) | 108.97 (11.54) | 102.30 (14.35)
  Shopping Trip 4 | 92.73 (10.76) | 116.16 (22.73) | 82.43 (9.38)
  Shopping Trip 5 | 73.07 (8.37) | 81.28 (9.48) | 82.46 (9.89)
  Shopping Trip 6 | 67.79 (8.40) | 70.37 (7.49) | 75.45 (9.29)

4. Secondary Outcome: Intensity Index for Cigarillos
Description: Number of cigarillos purchased at lowest price, averaged across the six shopping trips
Time Frame: Within the 20 minute survey.
Population: For this index, participants were removed whose baseline balance was insufficient to purchase any products and people who did not purchase anything. Another 50 cases were removed for violating modified bounce criterion.
Measure: Mean (Standard Deviation); unit: number of cigarillos
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 446 | 428 | 428
number of cigarillos | 6.33 (11.20) | 6.28 (9.75) | 6.64 (10.01)

5. Other Pre Specified Outcome: Negative Affect
Description: Three survey items to measure emotional reactions (anxious, scared, disgusted) to the cigarillo warning the participant saw. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 4 items and dividing by 4 (range 1-5), with higher scores representing a higher amount of the construct.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cognitive Elaboration
Description: The 1 item measure assesses the extent to which a participant reports the warning making them think about the risks of cigarillo smoking. Response options are on a 1 to 5 scale, with higher scores representing a higher amount of the construct.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Intentions to Quit Using Cigarillos
Description: Three survey items to measure participant's interest in quitting cigarillo smoking in the next month, likelihood of quitting smoking cigarillos in the month week, and plans to quit smoking cigarillos in the next month. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing the scores of the 3 items and dividing by 3 (range 1-5), with higher scores representing a higher amount of the construct/intentions to quit
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Warning Recall
Description: one survey item asking participants if they noticed any health warnings on the cigarillo packages during their shopping tasks, with response options of Yes, No, and I'm not sure. Recall will be determine if participants select Yes.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Warning Recognition
Description: One survey item asking participants to identify which warning they saw during their mock shopping trips. Participants will be shown their warning, a warning that wasn't in their ETM, and "I don't know" response options. Selecting the correct warning indicates warning recognition.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Perceived Message Effectiveness
Description: The 3-item UNC mean perceived message effectiveness scale assesses a participant's judgement of a warning's impact on their cigarillo beliefs and behavior. Response options are on a 1 to 5 scale. Overall scores are determined by summing the scores of the 3 items and dividing by 3 (range 1-5), with higher scores representing a higher amount of the construct
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Self-Reported Learning
Description: One survey item asking participants to what extent did they learn something new from the warning. Response options are on a 1 to 5 scale, with the higher number indicating more self-reported learning.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Average Total Amount of Non-tobacco Products Purchased
Description: Participants will participate in six mock shopping trips with a specified budget. They will have the option to purchase (mock) tobacco products in addition to cigarillos: cigarettes, menthol cigarettes, e-cigarettes/vaping devices, oral nicotine, and two non-tobacco options: snack food and non-alcoholic beverage. This outcome will be the sum mg of the number of non- tobacco products purchased during each of the six mock shopping trips.
Time Frame: Within the 20-minute survey
Reporting Status: Not Posted

13. Secondary Outcome: Cost Related Indices for Cigarillos
Description: Omax is the maximum amount spent on cigarillos across all shopping trips. Breakpoint is the price where no cigarillos were purchased. Pmax is the price where Omax occurs.
Time Frame: Within the 20-minute survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 446 | 428 | 428
dollars
  Omax-maximum amount spent across all shopping trips | 8.91 (10.46) | 9.89 (12.35) | 9.47 (11.10)
  Breakpoint-price where no cigarillos purchased | 6.05 (3.47) | 6.40 (3.27) | 6.37 (5.59)
  Pmax-price where Omax occurs | 3.05 (2.27) | 3.19 (2.26) | 3.04 (2.22)

14. Secondary Outcome: Rate of Change for Cigarillo Demand
Description: The rate of change for cigarillo demand is called Alpha, which is the rate constant of fitted Exponentiated Demand Equation. It is calculated with the Exponentiated Demand Equation, Q=Q0*10^k(e-αQ0C -1), where Q is the mg of nicotine purchased at a given price, Q0 is peak demand consumption or intensity (typically occurring at the lowest price), k is a constant across all compared conditions, and alpha (α) is the rate of change in demand or elasticity.
Time Frame: Within the 20-minute survey
Population: For Alpha, cases were removed for negative alphas values indicating poor/implausible fits. Cases were were also removed for negative curvature to the data (i.e., a mostly flat line), which does not allow alpha to be generated. Additional cases for each group were removed if alpha could not be calculated leading to the smaller numbers of participants analyzed in each group.
Measure: Mean (Standard Deviation); unit: cigarillos/dollar
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
Number analyzed (Participants) | 337 | 329 | 341
cigarillos/dollar | 0.03 (0.05) | 0.02 (0.03) | 0.03 (0.05)

ADVERSE EVENTS:
Time Frame: 20 minutes
Description: Study is minimal risk
Arm/Group | Cigarillo Warnings-Surgeon General Text-Only | Cigarillo Warnings-FDA Proposed Text-only | Cigarillo Warnings-Pictorial
All-Cause Mortality (participants affected / at risk) | 0/526 | 0/526 | 0/526
Serious Adverse Events (participants affected / at risk) | 0/526 | 0/526 | 0/526
Other Adverse Events (participants affected / at risk) | 0/526 | 0/526 | 0/526

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT05434013/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT05434013/ICF_000.pdf